CLINICAL TRIAL: NCT02578056
Title: Advanced Genital Prolapse Surgery With and Without Mid Urethral Sling to Prevent Stress Urinary Incontinence. A Multicenter, Randomized, Double-blind, Controlled Study
Brief Title: Advanced Genital Prolapse Surgery With and Without Mid Urethral Sling to Prevent Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Jorge Milhem Haddad, Head Chef of Urogynecology Section - University of Sao Paulo General Hospital, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IUOc
Record Dates: First submitted 2015-10-08; First posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Pelvic Organ Prolapse; Urinary Stress Incontinence
Keywords: pelvic organ prolapse; urinary incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress; Urinary Incontinence | interventions — Suburethral Slings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mid-urethral sling (Experimental): Patients randomized to anti-incontinence surgery will undergo TVT sling placement as the standard technique at the same time of genital prolapse surgery.
  Interventions: Device: Midurethral sling; Procedure: Genital prolapse surgery
- POP (Sham Comparator): Patients randomized to the sham group will be submitted to genital prolapse surgery and sham incisions as if they had undergone the TVT procedure (two small incisions of 0.5 cm in the suprapubic region in a similar way to that used for the insertion of the sling). These incisions intended to keep the raters blind to the achievement or otherwise of the sling during the postoperative evaluation.
  Interventions: Procedure: Genital prolapse surgery

INTERVENTIONS:
Device: Midurethral sling — Anti-urinary incontinence procedure, in a prophylactic way.
  Other Names: TVT Exact
  Arms: Mid-urethral sling
Procedure: Genital prolapse surgery — Surgical correction of genital prolapse

SUMMARY:
Pelvic organ prolapse (POP) is a public health problem worldwide, affecting about 30 %. It implies physical, psychological and social losses. A frequent complication after surgeries for POP is developing de novo stress urinary incontinence (SUI). SUI and POP have similar pathophysiology and therefore it is common to coexist in the same patient. De novo SUI has a prevalence 11-44 % after surgical correction of genital prolapse. Occult urinary incontinence (OUI) is considered the major risk factor for postoperative SUI. Studies on this topic show conflicting results. In a recent meta-analysis on this subject, Maher et al concluded that the value of performing any anti- incontinence procedure in continent women undergoing prolapse surgery remains unknown.

The aims of this study are to evaluate whether the association of a transvaginal tape (TVT®) in continent patients undergoing surgery for prolapse decreases the risk of de novo SUI and if it implies an improvement in their quality of life. The secondary endpoints are to assess the complications associated with this procedure, as irritative symptoms and voiding dysfunction postoperatively and assessing the ability of stress testing with reduced POP and urodynamics in predicting the risk of de novo SUI. This study will be a prospective, multicentric, randomized experimental study.

Patients with anterior or apical prolapse stages 3 and 4 (POP - Q) will be invited to participate in the study. The study will assess these patients for staging of prolapse, the presence of occult urinary incontinence and quality of life. Selected patients will be randomized to perform correction of genital prolapse and prophylactic anti-incontinence procedure or correction of genital prolapse only. Patients will be assessed 3, 6 and 12 months after surgery. Postoperative evaluation will be similar to preoperative. The exclusion criteria are: complaint or diagnosis of stress urinary incontinence before reduction of the prolapse, previous surgery for incontinence or pelvic organ prolapse, hypocontractility detrusor in urodynamics and inability to understand and give informed consent.

DETAILED DESCRIPTION:
The sample size calculation was based on a study with similar design. It was estimated that 312 patients would be sufficient to demonstrate a 15% difference between groups in a sample with 80% power and a significance level of 95 %. Considering a 20% margin of loss throughout the study we came to the final sample of 374 patients.

Preoperative evaluation: Genital prolapse will be staged according to the system of quantification of pelvic organ prolapse (ICS Pelvic Organ Quantification Prolapse - POP - Q ). All patients will be initially analyzed for quantitative urinalysis and urine culture prior to testing to IUO. In case of urinary infection, the patient will be subjected to antibiotics and reassessed after a negative urine culture. To perform the effort test, during the physical examination, the patient's bladder will be emptied with a urinary catheter and soon after instilled with 300ml of saline solution. By this time the stress test (Valsalva maneuver and cough) will be held before and after prolapse reduction. The test will be performed with the patient in supine and prone positions. The prolapse reduction will be performed using gauzes on a DeLee forceps. The urodynamics consists of three stages: initial uroflowmetry, cystometry and voiding study. The stress test will be performed during cystometry in the cystometric capacity of 300ml, with and without prolapse reduction. The reduction will be carried out on the same fashion as stress test. Schafer nomogram will be used for the diagnosis of detrusor hypocontractility and the Blaivas - Groutz nomogram for the diagnosis of obstruction. The presence of urinary incontinence after prolapse reduction in the clinical stress test or urodynamics configure the diagnosis of occult stress urinary incontinence.

The patients will be submitted for assessment of quality of life through the following questionnaires : Quality of Life Questionnaire Prolapse and Incontinence Quality of Life Questionnaire ( I-QOL ).

The surgical repair will be conducted on this way: Surgical correction of genital prolapse will be taken vaginally. The prolapse of the anterior vaginal wall will be treated with site-specific correction of pubocervical fascia . The correction of apical prolapse will be performed with the use of High McCall culdoplasty technique. In uterine prolapse, associated vaginal hysterectomy will be performed.

The posterior vaginal wall prolapse will be treated with site-specific correction of rectovaginal fascia.If present, the perineal tear will be corrected.

Patients randomized to anti-incontinence surgery will undergo TVT as standard technique. Patients randomized to pelvic organ prolapse surgery alone will undergo two small incisions of 0.5 cm in the suprapubic region in a similar way to that used for the insertion of the sling (sham incisions). These incisions intended to keep the raters blind to the achievement or otherwise of the sling during the postoperative evaluation.

Randomization will be held by a computer-generated random numbers software. The result of randomization will be revealed in the operating room after the patient is anesthetized, ie, the patient will be blinded for carrying or not a sling. The surgeon will be blinded to the results of preoperative IUO evaluation and results of quality of life questionnaires. Patients and researchers who will carry out the postoperative evaluations will be blinded to treatment.

Statistical Evaluation Continuous variables will be presented as mean and standard deviation and compared using the two-tailed Student t test for two samples. Categorical variables will be presented as frequencies and percentages and compared between groups by the Fisher exact test, p < 0.05 will be considered statistically significant. These evaluations will be performed using a SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* genital prolapse POP-Q stages 3 or 4
* surgical treatment planning.

Exclusion Criteria:

* signals or symphtoms of stress urinary incontinence before prolapse reduction
* previous surgery for stress urinary incontinence
* previous surgery for genital prolapse
* inability to understand and give informed consent

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2014-02; Primary Completion 2020-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of de novo stress urinary incontinence | 3, 6 and 12 months postoperatively
  Number of participants presenting with de novo stress urinary incontinence as assessed by simple clinical examination (3 and 12 months) or with an standadized effort test (6m) and by the Incontinence Quality of Life Questionnaire (not answering NO to the question number 2).

SECONDARY OUTCOMES:
Complications related to the surgical procedure (s) | 7 days postoperatively
  Number of participants with intra-operative complications, such as hemorrhage and organ damage (bladder, urethral or intestinal). Intraoperative bleeding will be evaluated subjectively by the surgeons by answering the following question: There was an hemorrhage during the surgical procedure? ( ) Yes ( )No. Did the patient need to get a blood transfusion? ( ) No ( ) Yes: number of packed red blood cells transfunded ____.
  Organ damage will be reported by the surgeon on the perioperative record by answering the question. Were there complications as organ damage during the surgery? ( ) No ( ) Yes: ( ) Bladder injury ( ) Urethra injury ( ) Intestinal Injury
Incidence of overactive bladder and urinary obstruction symptoms | 3, 6 and 12 months postoperatively
  Number of participants with overactive bladder and/or urinary obstruction symptoms as assessed by the Incontinence Quality of Life Questionnaire (questions numbers 1,3, 4 and 10) and the Prolapse Quality of Life Questionnaire (Questions 3, 4, 5 and 6).
Positive predictive value of urodynamics and Standadized Effort Test to detect patients who will became incontinence after surgery. | 3, 6 and 12 months postoperatively
  The investigators will calculate the ability of urodinamics and stardadized effort test to predict postoperative stress urinary incontinece in the sham group. For this purpouse the positive predictive value of each test will be calculated.
Negative predictive value of urodynamics and Standadized Effort Test to detect patients who will remain continents after surgery. | 3, 6 and 12 months
  The investigators will calculate the ability of urodinamics and stardadized effort test to predict postoperative continent patients in the sham group. For this purpouse the negative predictive value os each test will be calculated.
Impact of urinary incontinence on patient´s quality of life | 3, 6 and 12 months
  Average score in the Incontinence Quality of Life Questionnaire on each group
Impact of prolapse on patient´s quality of life | 12 months
  average score in the prolapse quality of life questionnaire
need for surgery or any treatment for urinary incontinence postoperatively | 12 months
  The investigators will evaluate the number of patients that requested addicional treatment for urinary incontinence 12 months after the inicial surgery, on each group.
Eficaccy of surgery to treat and relief prolapse symptoms | 12 months
  The investigators will evaluate the eficcacy of the proposed surgical technic for the treatment of genital prolapse as assessed by symptoms (Prolapse Quality of Life Questionnaire) and the POP-Q classification on physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana p gomes, MD, Principal Investigator — University of Sao Paulo Medical School
Locations (1):
- University of sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Swift SE. The distribution of pelvic organ support in a population of female subjects seen for routine gynecologic health care. Am J Obstet Gynecol. 2000 Aug;183(2):277-85. doi: 10.1067/mob.2000.107583. PMID 10942459
- [Background] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Background] Malak M. The role of anti-incontinence surgery in management of occult urinary stress incontinence. Int Urogynecol J. 2012 Jul;23(7):823-5. doi: 10.1007/s00192-011-1563-4. Epub 2011 Sep 17. PMID 21927940
- [Background] Brubaker L, Nygaard I, Richter HE, Visco A, Weber AM, Cundiff GW, Fine P, Ghetti C, Brown MB. Two-year outcomes after sacrocolpopexy with and without burch to prevent stress urinary incontinence. Obstet Gynecol. 2008 Jul;112(1):49-55. doi: 10.1097/AOG.0b013e3181778d2a. PMID 18591307
- [Background] Wei JT, Nygaard I, Richter HE, Nager CW, Barber MD, Kenton K, Amundsen CL, Schaffer J, Meikle SF, Spino C; Pelvic Floor Disorders Network. A midurethral sling to reduce incontinence after vaginal prolapse repair. N Engl J Med. 2012 Jun 21;366(25):2358-67. doi: 10.1056/NEJMoa1111967. PMID 22716974
- [Background] Maher CM, Feiner B, Baessler K, Glazener CM. Surgical management of pelvic organ prolapse in women: the updated summary version Cochrane review. Int Urogynecol J. 2011 Nov;22(11):1445-57. doi: 10.1007/s00192-011-1542-9. Epub 2011 Sep 17. PMID 21927941
- [Background] Stanton SL, Hilton P, Norton C, Cardozo L. Clinical and urodynamic effects of anterior colporrhaphy and vaginal hysterectomy for prolapse with and without incontinence. Br J Obstet Gynaecol. 1982 Jun;89(6):459-63. doi: 10.1111/j.1471-0528.1982.tb03637.x. PMID 7082603
- [Background] Schierlitz L, Dwyer PL, Rosamilia A, De Souza A, Murray C, Thomas E, Hiscock R, Achtari C. Pelvic organ prolapse surgery with and without tension-free vaginal tape in women with occult or asymptomatic urodynamic stress incontinence: a randomised controlled trial. Int Urogynecol J. 2014 Jan;25(1):33-40. doi: 10.1007/s00192-013-2150-7. Epub 2013 Jun 28. PMID 23812579
- [Background] Souza CC, Rodrigues AM, Ferreira CE, Fonseca ES, di Bella ZI, Girao MJ, Sartori MG, Castro RA. Portuguese validation of the Urinary Incontinence-Specific Quality-of-Life Instrument: I-QOL. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Oct;20(10):1183-9. doi: 10.1007/s00192-009-0916-8. Epub 2009 Jun 9. PMID 19506791
- [Background] de Oliveira MS, Tamanini JT, de Aguiar Cavalcanti G. Validation of the Prolapse Quality-of-Life Questionnaire (P-QoL) in Portuguese version in Brazilian women. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Oct;20(10):1191-202. doi: 10.1007/s00192-009-0934-6. Epub 2009 Jul 4. PMID 19578803